CLINICAL TRIAL: NCT01325805
Title: Pregnancy Outcomes in Overweight and Obese Women With a History of Recurrent Pregnancy Loss Randomized to a Structured Weight Loss Program Versus Routine Weight-Loss Counseling: A Pilot Study
Brief Title: Efficacy of a Structured Weight Loss Program in Overweight Women With a History of Recurrent Pregnancy Loss
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult to recruit, very poor compliance with interventions
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Ruth Bunker Lathi, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-03212011-7603; IRB Protocol Number 20001 (Other: Stanford University)
Record Dates: First submitted 2011-03-23; First posted 2011-03-30 (Estimated); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Obese; Overweight; Miscarriage; Recurrent Pregnancy Loss
Keywords: Miscarriage; Recurrent Pregnancy Loss; Obesity; Overweight; Diet
MeSH Terms: conditions — Obesity; Overweight; Abortion, Spontaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Structured Weight Loss (Experimental): Women randomized to this arm will meet with a registered dietician regularly for review of calorie recommendations and food diary. As well as regular clinic visits to measure patients weight.
  Interventions: Behavioral: Structured Weight Loss Program
- Routine Weight Loss Counseling (Active Comparator): Patients are counseled by a physicians about the impact of maternal weight on fertility and pregnancy outcomes.
  Interventions: Behavioral: Routine Weight Loss Counseling

INTERVENTIONS:
Behavioral: Structured Weight Loss Program — Those patients randomized to the structured weight loss group will have a formal evaluation and counseling a medical endocrinologist specializing in weight management. The structured weight loss program will consist of meeting with a dietician who will guide them on following a hypocaloric diet with a calorie deficit of 750kcal/day. The weight loss goal will be to lose 1-1.5 pounds/week. The participants will receive teaching utilizing the American Diabetes Association Exchange Lists and will receive sample meal plans. In addition, participants will be seen by the dietitian once a week for a month, then every 2 weeks for 2 months, then once per month for 3 months. Patients randomized to the study group will continue in the structured weight loss program for 6 months.
  Arms: Structured Weight Loss
Behavioral: Routine Weight Loss Counseling — Participants randomized to the routine weight loss counseling group will receive the ACOG Patient Education pamphlets on obesity.
  Arms: Routine Weight Loss Counseling

SUMMARY:
Overweight and obesity has been associated with a number of adverse pregnancy outcomes in women of reproductive age, including infertility and early pregnancy loss. Recent data suggests that overweight and obese patients are also at increased risk of recurrent pregnancy loss (RPL), a devastating condition that affects 1% of the fertile population.

The investigators propose a prospective, randomized controlled trial in which overweight and obese patients with unexplained recurrent pregnancy loss are enrolled in a structured, 6 month, weight loss program or provided routine counseling regarding the importance of weight loss. Pregnancy outcomes will then be followed to assess miscarriage rates. Metabolic outcomes, such as lipid and glucose profiles, will also be evaluated.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the impact of a structured weight loss program versus traditional weight-loss counseling on pregnancy outcomes in women with recurrent pregnancy loss. The study protocol is as follows:

1. Patients will be notified of study via flyer inserted into patient chart at initial clinic visit, physician referral or Stanford website. Patients expressing interest will have their charts reviewed to confirm that they meet all enrollment criteria. Potential subjects will then be contacted via phone and verbal consent to participate obtained.
2. The participant will then have an office visit for consent signing and randomization. A formal weight will be obtained, the Beck Depression Inventory will be administered by Penny Donnelly, a self-administered questionnaire will be completed, and a basic laboratory evaluation, including a fasting lipid panel, alanine aminotransferase (ALT), fasting glucose and insulin levels, 2-hour glucose tolerance test, hemoglobin A1c and CRP will be preformed.
3. The patients will then be randomized to traditional weight loss counseling (control group) or to the structured weight loss program (study group). Patients will be instructed to discontinue attempts at conception.
4. Those patients randomized to the control group will receive the ACOG Patient Education pamphlets on obesity.
5. Those patients randomized to the study group will have a formal evaluation and counseling by Dr. Sun Kim, a medical endocrinologist specializing in weight management. They will then be enrolled in a structured weight loss program.
6. For all patients, a 3-month follow-up office visit will be scheduled. At this visit, a formal weight will be obtained, the Beck Depression Inventory will be re-administered by Penny Donnelly, a self-administered questionnaire will be completed, and a follow-up laboratory evaluation, including a fasting lipid panel, alanine aminotransferase (ALT), fasting glucose and insulin levels, 2-hour glucose tolerance test, hemoglobin A1c and CRP will be preformed. Patients will be informed that they may now being attempts to conceive.
7. Patients randomized to the study group will continue in the structured weight loss program for 6 months.
8. Six months after enrollment, all patients will have a telephone interview in which a close-out questionnaire will be administered and a final, self-reported weight will be obtained.
9. Primary and secondary outcomes will be followed for 2.5 years after date of enrollment for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Unexplained recurrent pregnancy loss (2 or more prior miscarriages)
2. BMI >=25 kg/m2
3. Prepared to take 3 months ¡®time out¡± from attempting to conceive
4. Ability to attend a one hour initial, then 30 minute follow-up nutrition/monitoring session - once per week for one month, then every other week for 2 months, then once then once per month for 3 months.

Exclusion Criteria:

1. Age >=40 years
2. Diagnosis of Type 1 or Type 2 Diabetes as defined by a fasting glucose >=126, or 2 hour glucose >=200 by a 75 gram oral glucose challenge
3. Presence of an endocrine condition such as hyperprolactinemia, Cushing¡-s syndrome or untreated thyroid disease (defined as a TSH outside of the laboratory determined normal range)
4. Desire to continue attempts to conceive for the duration of the program
5. History of bariatric surgery
6. Use of over-the-counter or prescribed weight loss medications with the exception of metformin
7. Enrollment in another clinical trial (excluding surveys)

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Term live birth rate | 2.5 years

SECONDARY OUTCOMES:
Weight loss - goal for weight loss defined as 5 percent of enrollment body weight lost | 6 months
Changes in triglyceride levels | 3 months
Changes in high density lipoprotein levels | 3 months
Changes in alanine aminotransferase (ALT) levels | 3 months
Changes in fasting insulin levels | 3 months
Changes in postprandial insulin levels | 3 months
Changes in fasting glucose levels | 3 months
Changes in postprandial glucose levels | 3 months
Changes in hemoglobin A1c levels | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Bunker Lathi, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Practice Committee of tAmerican Society for Reproductive Medicine. Definitions of infertility and recurrent pregnancy loss. Fertil Steril. 2008 Nov;90(5 Suppl):S60. doi: 10.1016/j.fertnstert.2008.08.065. PMID 19007647
- [Background] Li TC, Makris M, Tomsu M, Tuckerman E, Laird S. Recurrent miscarriage: aetiology, management and prognosis. Hum Reprod Update. 2002 Sep-Oct;8(5):463-81. doi: 10.1093/humupd/8.5.463. PMID 12398226
- [Background] James PT. Obesity: the worldwide epidemic. Clin Dermatol. 2004 Jul-Aug;22(4):276-80. doi: 10.1016/j.clindermatol.2004.01.010. PMID 15475226
- [Background] Shirazian T, Raghavan S. Obesity and pregnancy: implications and management strategies for providers. Mt Sinai J Med. 2009 Dec;76(6):539-45. doi: 10.1002/msj.20148. PMID 20014418
- [Background] Rich-Edwards JW, Goldman MB, Willett WC, Hunter DJ, Stampfer MJ, Colditz GA, Manson JE. Adolescent body mass index and infertility caused by ovulatory disorder. Am J Obstet Gynecol. 1994 Jul;171(1):171-7. doi: 10.1016/0002-9378(94)90465-0. PMID 8030695
- [Background] Jensen MD. Medical management of obesity. Semin Gastrointest Dis. 1998 Oct;9(4):156-62. PMID 9822077
- [Background] Bolumar F, Olsen J, Rebagliato M, Saez-Lloret I, Bisanti L. Body mass index and delayed conception: a European Multicenter Study on Infertility and Subfecundity. Am J Epidemiol. 2000 Jun 1;151(11):1072-9. doi: 10.1093/oxfordjournals.aje.a010150. PMID 10873131
- [Background] van der Steeg JW, Steures P, Eijkemans MJ, Habbema JD, Hompes PG, Burggraaff JM, Oosterhuis GJ, Bossuyt PM, van der Veen F, Mol BW. Obesity affects spontaneous pregnancy chances in subfertile, ovulatory women. Hum Reprod. 2008 Feb;23(2):324-8. doi: 10.1093/humrep/dem371. Epub 2007 Dec 11. PMID 18077317
- [Background] Metwally M, Ong KJ, Ledger WL, Li TC. Does high body mass index increase the risk of miscarriage after spontaneous and assisted conception? A meta-analysis of the evidence. Fertil Steril. 2008 Sep;90(3):714-26. doi: 10.1016/j.fertnstert.2007.07.1290. Epub 2008 Feb 6. PMID 18068166
- [Background] Lashen H, Fear K, Sturdee DW. Obesity is associated with increased risk of first trimester and recurrent miscarriage: matched case-control study. Hum Reprod. 2004 Jul;19(7):1644-6. doi: 10.1093/humrep/deh277. Epub 2004 May 13. PMID 15142995
- [Background] Wang JX, Davies MJ, Norman RJ. Obesity increases the risk of spontaneous abortion during infertility treatment. Obes Res. 2002 Jun;10(6):551-4. doi: 10.1038/oby.2002.74. PMID 12055331
- [Background] Metwally M, Saravelos SH, Ledger WL, Li TC. Body mass index and risk of miscarriage in women with recurrent miscarriage. Fertil Steril. 2010 Jun;94(1):290-5. doi: 10.1016/j.fertnstert.2009.03.021. Epub 2009 May 12. PMID 19439294
- [Background] Clark AM, Thornley B, Tomlinson L, Galletley C, Norman RJ. Weight loss in obese infertile women results in improvement in reproductive outcome for all forms of fertility treatment. Hum Reprod. 1998 Jun;13(6):1502-5. doi: 10.1093/humrep/13.6.1502. PMID 9688382
- See also: Stanford Fertility & Reproductive Medicine Center — https://fertility.stanfordchildrens.org